CLINICAL TRIAL: NCT00955409
Title: A PHASE IIA, MULTICENTER, RANDOMIZED, THIRD-PARTY UNBLINDED, LONG -TERM EXTENSION STUDY TO DETERMINE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF ACC-001 WITH QS-21 ADJUVANT IN SUBJECTS WITH MILD TO MODERATE ALZHEIMER'S DISEASE
Brief Title: Long Term Extension Study Evaluating Safety, Tolerability and Immunogenicity Of ACC-001 In Subjects With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3134K1-2203; B2571007 (Other: Alias Study Number); 2009-010922-21 (EudraCT Number)
Record Dates: First submitted 2009-08-04; First posted 2009-08-10 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — vanutide cridificar; saponin QA-21V1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ACC-001(3µg) + QS21 (Experimental): ACC-001(3µg) + QS21
  Interventions: Biological: ACC-001(3µg) + QS21
- ACC-001(10µg) + QS21 (Experimental): ACC-001(10µg) + QS21
  Interventions: Biological: ACC-001(10µg) + QS21
- ACC-001(30µg) + QS21 (Experimental): ACC-001(30µg) + QS21
  Interventions: Biological: ACC-001(30µg) + QS21

INTERVENTIONS:
Biological: ACC-001(3µg) + QS21 — Vanutide Cridificar (ACC-001) 3µg + QS-21 (50µg), IM on Day 1, Month 6, Month 12 and Month 18
  Arms: ACC-001(3µg) + QS21
Biological: ACC-001(10µg) + QS21 — Vanutide Cridificar (ACC-001) 10µg + QS-21 (50µg), IM on Day 1, Month 6, Month 12 and Month 18
  Arms: ACC-001(10µg) + QS21
Biological: ACC-001(30µg) + QS21 — Vanutide Cridificar (ACC-001) 30 µg + QS-21 (50µg), IM on Day 1, Month 6, Month 12 and Month 18
  Arms: ACC-001(30µg) + QS21

SUMMARY:
The purpose of this study is to assess the long term safety, tolerability, and immunogenicity of ACC-001, an investigational active immunization product+, in subjects with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects randomized under previous 3134K1-200 study (NCT00479557) and met all inclusion/and none of the exclusion criteria
* Screening brain MRI scan is consistent with the diagnosis of AD ' Mini-Mental State Examination (MMSE) score ≥10

Exclusion Criteria:

* Significant Neurological Disease other than Alzheimer's disease
* Brain MRI evidence of vasogenic edema (VE) during the preceding 3134K1 200 study (NCT00479557)
* Clinically significant systemic illness

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-11-05 (Actual); Primary Completion 2013-12-17 (Actual); Study Completion 2013-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- France (8):
  - CMRR Bordeaux CHU Pellegrin, Bordeaux
  - Hopital Roger Salengro, Lille
  - Hôpital Roger Salengro, Lille
  - CHU La Timone, Marseille
  - Groupe Hospitalier Broca-La Rochefoucauld, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - Hôpital La Grave, Toulouse
- Germany (6):
  - Klinik fuer Psychiatrie und Psychotherapie, Charite Universitaetsmedizin Berlin, Berlin
  - Universitatsklinikum und Poliklinik der Uni Bonn, Bonn
  - Klinikum der Albert-Ludwigs-Universitaet Freiburg, Freiburg im Breisgau
  - Klinik fuer Psychiatrie und Psychotherapie, Göttingen
  - Zentralinstitut fuer Seelische Gesundheit Mannheim, Mannheim
  - Technische Universität München, Munich
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinico y Provincial, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3134K1-2203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned duration was approximately 2 years (including 18 months of treatment + 6 months of follow-up). Participants who completed the lead-in 3134K1-200-EU (B2571004) study through Week 78 (Week 104 for Cohort 1 and 2) had the option to stay in the lead-in study or to roll-over into the extension protocol 3134K1-2203-EU (B2571007).
Pre-assignment Details: The Basic Results disclose pooled data from the extension studies 3134K1-2203-EU (B2571007) and 3134K1-2205-US (B2571008).
Groups:
- ACC 3 µg+QS-21 / ACC 3 µg+QS-21: Participants received 3 μg of ACC-001 and 50 μg of QS-21 in the lead-in study and in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- QS-21 / ACC 3 µg+QS-21: Participants received 50 μg of QS-21 in the lead-in study and 3 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- ACC 10 µg+QS-21 / ACC 10 µg+QS-21: Participants received 10 μg of ACC-001 and 50 μg of QS-21 in the lead-in study and in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- ACC 10 µg / ACC 10 µg+QS-21: Participants received 10 μg of ACC-001 in the lead-in study and 10 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- QS-21 / ACC 10 µg+QS-21: Participants received 50 μg of QS-21 in the lead-in study and 10 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- PBS / ACC 10 µg+QS-21: Participants received Phosphate buffered Saline (PBS) in the lead-in study and 10 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- ACC 30 µg+QS-21 / ACC 30 µg+QS-21: Participants received 30 μg of ACC-001 and 50 μg of QS-21 in the lead-in study and in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- ACC 30 µg / ACC 30 µg+QS-21: Participants received 30 μg of ACC-001 in the lead-in study and 30 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- QS-21 / ACC 30 µg+QS-21: Participants received 50 μg of QS-21 in the lead-in study and 30 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- PBS / ACC 30 μg+QS-21: Participants received PBS in the lead-in study and 30 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
Period: Overall Study
Arm/Group | ACC 3 µg+QS-21 / ACC 3 µg+QS-21 | QS-21 / ACC 3 µg+QS-21 | ACC 10 µg+QS-21 / ACC 10 µg+QS-21 | ACC 10 µg / ACC 10 µg+QS-21 | QS-21 / ACC 10 µg+QS-21 | PBS / ACC 10 µg+QS-21 | ACC 30 µg+QS-21 / ACC 30 µg+QS-21 | ACC 30 µg / ACC 30 µg+QS-21 | QS-21 / ACC 30 µg+QS-21 | PBS / ACC 30 μg+QS-21
Started | 21 (Started=Randomized) | 6 (Started=Randomized) | 41 (Started=Randomized) | 25 (Started=Randomized.) | 5 (Started=Randomized) | 9 (Started=Randomized) | 27 (Started=Randomized) | 6 (Started=Randomized) | 16 (Started=Randomized) | 4 (Started=Randomized)
Treated | 21 | 6 | 41 | 24 | 5 | 9 | 27 | 6 | 16 | 4
Completed Treatment | 12 | 5 | 15 | 17 | 3 | 7 | 4 | 3 | 2 | 4
Completed | 11 (Completed study) | 5 (Completed study) | 15 (Completed study) | 17 (Completed study) | 3 (Completed study) | 6 (Completed study) | 3 (Completed study) | 2 (Completed study) | 2 (Completed study) | 3 (Completed study)
Not Completed | 10 | 1 | 26 | 8 | 2 | 3 | 24 | 4 | 14 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 5 | 2 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Caregiver Request | 2 | 0 | 6 | 5 | 0 | 2 | 3 | 1 | 3 | 0
Not completed — Investigator Request | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Discontinuation of Study by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Failed to Return | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event (AE) | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0
Not completed — Reason not Specified | 2 | 1 | 13 | 1 | 2 | 0 | 16 | 0 | 8 | 1

BASELINE CHARACTERISTICS:
Population: 160 participants were randomized and included in analysis. Of these, 1 participant was not treated: at screening, the site felt that Mini-Mental State Examination (MMSE) score was artificially low due to language issue. Hence, study enrollment was approved. Later, participant discontinued from study, which was recorded as major protocol deviation.
Groups:
- PBS / ACC 10 μg+QS-21: Participants received PBS in the lead-in study and 10 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- Total: Total of all reporting groups
Arm/Group | ACC 3 µg+QS-21 / ACC 3 µg+QS-21 | QS-21 / ACC 3 µg+QS-21 | ACC 10 µg+QS-21 / ACC 10 µg+QS-21 | ACC 10 µg / ACC 10 µg+QS-21 | QS-21 / ACC 10 µg+QS-21 | PBS / ACC 10 μg+QS-21 | ACC 30 µg+QS-21 / ACC 30 µg+QS-21 | ACC 30 µg / ACC 30 µg+QS-21 | QS-21 / ACC 30 µg+QS-21 | PBS / ACC 30 μg+QS-21 | Total
Number analyzed (Participants) | 21 | 6 | 41 | 25 | 5 | 9 | 27 | 6 | 16 | 4 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (6.94) | 67.7 (9.52) | 69.7 (9.29) | 72.4 (9.12) | 75.2 (8.23) | 69.6 (7.94) | 71.3 (9.20) | 66.3 (9.42) | 69.5 (6.95) | 75.8 (7.89) | 70.4 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 21 | 12 | 3 | 8 | 16 | 3 | 14 | 2 | 94
  Male | 10 | 2 | 20 | 13 | 2 | 1 | 11 | 3 | 2 | 2 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
  Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 20 | 6 | 40 | 25 | 4 | 9 | 26 | 6 | 16 | 4 | 156
MMSE Score [Mean (Standard Deviation); unit: score] — The Mini Mental Score Examination (MMSE) is a clinical instrument used for detecting cognitive impairment of the participants and assessing its severity. It is a brief, structured 11 item questionnaire that tests 5 areas of cognitive function: orientation, registration, attention and calculation, recall and language. The total score ranges from 0 to 30 and the following cut off was used for MMSE ranges >26 = no impairment; 21-26 = mild impairment; 10-20 = moderate impairment; <10 = severe impairment.
  score | 16.7 (4.64) | 18.3 (5.61) | 18.4 (5.92) | 19.6 (5.45) | 21.8 (4.21) | 20.0 (6.14) | 18.7 (4.98) | 20.5 (4.76) | 19.1 (4.84) | 20.0 (4.69) | 18.8 (5.29)
MMSE Ranges [Count of Participants; unit: Participants]
  MMSE score >26 | 0 | 0 | 5 | 3 | 1 | 1 | 1 | 0 | 1 | 0 | 12
  MMSE score 21-26 | 5 | 2 | 9 | 7 | 2 | 3 | 8 | 3 | 6 | 3 | 48
  MMSE score 16-20 | 5 | 2 | 12 | 10 | 2 | 3 | 11 | 2 | 6 | 0 | 53
  MMSE score 10-15 | 10 | 2 | 15 | 5 | 0 | 2 | 7 | 1 | 3 | 1 | 46
  MMSE score <10 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Other Pre Specified Outcome: GMTs of Anti-A-beta Immunoglobulin M (IgM) Using ELISA at Weeks 0, 4, 12, 24, 30, 36, 50, 56, 66, 76, 82, and 104
Description: IGM was not statistically analyzed.
Time Frame: Weeks 0, 4, 12, 24, 30, 36, 50, 56, 66, 76, 82, and 104
Groups:
- ACC 10 µg+QS-21 / ACC 10 µg+QS-21: Participants 10 μg of ACC-001 and 50 μg of QS-21 in the lead-in study and in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- ACC 30 μg+QS-21 / ACC 30 μg+QS-21: Participants received 30 μg of ACC-001 and 50 μg of QS-21 in the lead-in study and in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- ACC 30 μg / ACC 30 μg+QS-21: Participants received 30 μg of ACC-001 in the lead-in study and 30 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- QS-21 / ACC 30 μg+QS-21: Participants received 50 μg of QS-21 in the lead-in study and 30 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
Arm/Group | ACC 3 µg+QS-21 / ACC 3 µg+QS-21 | QS-21 / ACC 3 µg+QS-21 | ACC 10 µg+QS-21 / ACC 10 µg+QS-21 | ACC 10 µg / ACC 10 µg+QS-21 | QS-21 / ACC 10 µg+QS-21 | PBS / ACC 10 μg+QS-21 | ACC 30 μg+QS-21 / ACC 30 μg+QS-21 | ACC 30 μg / ACC 30 μg+QS-21 | QS-21 / ACC 30 μg+QS-21 | PBS / ACC 30 μg+QS-21
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Other Pre Specified Outcome: Change From Baseline GMTs of Anti-A-beta IgG Subtypes Using ELISA at Visits Where an IgG Total Response is Measurable (at Weeks 0, 4, 12, 24, 30, 36, 50, 56, 66, 76, 82, and 104 if Applicable)
Description: IgG subtypes were not assessed
Time Frame: Weeks 0, 4, 12, 24, 30, 36, 50, 56, 66, 76, 82, and 104
Arm/Group | ACC 3 µg+QS-21 / ACC 3 µg+QS-21 | QS-21 / ACC 3 µg+QS-21 | ACC 10 µg+QS-21 / ACC 10 µg+QS-21 | ACC 10 µg / ACC 10 µg+QS-21 | QS-21 / ACC 10 µg+QS-21 | PBS / ACC 10 μg+QS-21 | ACC 30 μg+QS-21 / ACC 30 μg+QS-21 | ACC 30 μg / ACC 30 μg+QS-21 | QS-21 / ACC 30 μg+QS-21 | PBS / ACC 30 μg+QS-21
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Treatment-emergent AEs or Serious Adverse Events (SAEs)
Description: An AE was any untoward, undesired, or unplanned clinical event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given study drug or in a sponsor's clinical study. The event did not need to be causally related to the study drug or the clinical studies. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: 24 months
Population: All participants who received at least one dose of the study drug were included in the safety population. For safety analyses, the participants were summarized according to the combination of treatments they actually received during the 3134K1-200-EU or 3134K1-2201-US lead-in studies and 3134K1-2203-EU or 3134K1-2205-US extension studies.
Measure: Number; unit: percentage of participants
Groups:
- Active / ACC 10 µg+QS-21: Participants 10 μg of ACC-001 and 50 μg of QS-21 or 10 μg of ACC-001 alone in the lead-in study and 10 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- Control / ACC 10 µg+QS-21: Participants received 50 μg of QS-21 or PBS in the lead-in study and 10 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- Active / ACC 30 µg+QS-21: Participants received 30 μg of ACC-001 and 50 μg of QS-21 or 30 μg of ACC-001 alone in the lead-in study and 30 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- Control / ACC 30 μg+QS-21: Participants received 50 μg of QS-21 or PBS in the lead-in study and 30 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
Arm/Group | ACC 3 µg+QS-21 / ACC 3 µg+QS-21 | QS-21 / ACC 3 µg+QS-21 | Active / ACC 10 µg+QS-21 | Control / ACC 10 µg+QS-21 | Active / ACC 30 µg+QS-21 | Control / ACC 30 μg+QS-21
Number analyzed (Participants) | 21 | 6 | 65 | 14 | 33 | 20
percentage of participants
  Percentage of participants with AEs | 100.0 | 100.0 | 93.8 | 92.9 | 78.8 | 90.0
  Percentage of participants with SAEs | 28.6 | 0 | 24.6 | 14.3 | 12.1 | 20.0

4. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Anti-A-beta Immunoglobulin G (IgG) Total Using an Enzyme-linked Immunosorbent Assay (ELISA) at Weeks 0, 4, 12, 24, 30, 36, 50, 56, 66, 76, 82, and 104
Description: The lower limit of quantification (LLOQ) was 100 U/mL and when the assay result was below LLOQ (100 U/mL), 50 U/mL was imputed for IgG.
Time Frame: Weeks 0, 4, 12, 24, 30, 36, 50, 56, 66, 76, 82, and 104
Population: The immunogenicity population included all randomized participants with documented injection of at least one dose of study drug and at least one immunogenicity data point collected.
Measure: Geometric Mean (95% Confidence Interval); unit: U/ml
Arm/Group | ACC 3 µg+QS-21 / ACC 3 µg+QS-21 | QS-21 / ACC 3 µg+QS-21 | ACC 10 µg+QS-21 / ACC 10 µg+QS-21 | ACC 10 µg / ACC 10 µg+QS-21 | QS-21 / ACC 10 µg+QS-21 | PBS / ACC 10 μg+QS-21 | ACC 30 µg+QS-21 / ACC 30 µg+QS-21 | ACC 30 µg / ACC 30 µg+QS-21 | QS-21 / ACC 30 µg+QS-21 | PBS / ACC 30 μg+QS-21
Number analyzed (Participants) | 21 | 6 | 41 | 24 | 5 | 9 | 27 | 6 | 16 | 4
U/ml
  Screening Lead-in (N:21,6,41,24,5,9,27,6,16,4) | 50.0 [NA to NA] — Below level of detection | 50.0 [NA to NA] — Below level of detection | 50.0 [NA to NA] — Below level of detection | 50.0 [NA to NA] — Below level of detection | 50.0 [NA to NA] — Below level of detection | 50.0 [NA to NA] — Below level of detection | 50.0 [NA to NA] — Below level of detection | 50.0 [NA to NA] — Below level of detection | 58.8 [41.6 to 83.3] | 50.0 [NA to NA] — Below level of detection
  Screening Extension (N:21,6,41,24,5,9,27,6,16,4) | 836.5 [362.2 to 1932.3] | 50.0 [NA to NA] — Below level of detection | 1623.4 [1015.3 to 2595.7] | 180.2 [76.4 to 425.3] | 50.0 [NA to NA] — Below level of detection | 50.0 [NA to NA] — Below level of detection | 1718.3 [1101.2 to 2681.3] | 424.2 [70.9 to 2539.4] | 59.5 [41.0 to 86.3] | 50.0 [NA to NA] — Below level of detection
  Week 4 (N:21,6,41,24,5,9,27,5,16,4) | 4523.7 [2070.2 to 9885.0] | 50.0 [NA to NA] — Below level of detection | 6219.3 [3853.2 to 10038.2] | 517.9 [166.8 to 1607.6] | 50.0 [NA to NA] — Below level of detection | 60.6 [38.9 to 94.4] | 8436.2 [5569.8 to 12778.0] | 4223.0 [185.0 to 96408.3] | 144.7 [67.9 to 308.0] | 100.1 [11.0 to 912.6]
  Week 12 (N:21,6,41,23,4,9,27,5,16,4) | 2540.3 [1060.5 to 6084.8] | 50.0 [NA to NA] — Below level of detection | 4251.0 [2709.7 to 6669.2] | 425.4 [137.0 to 1320.6] | 50.0 [NA to NA] — Below level of detection | 62.0 [37.8 to 101.7] | 3604.3 [2009.6 to 6464.5] | 761.6 [33.2 to 17472.9] | 89.3 [43.7 to 182.5] | 87.9 [14.6 to 529.8]
  Week 24 (N:21,6,39,24,4,9,27,5,15,3) | 1466.6 [607.2 to 3542.4] | 50.0 [NA to NA] — Below level of detection | 3058.1 [1887.1 to 4955.9] | 280.3 [100.2 to 784.4] | 50.0 [NA to NA] — Below level of detection | 57.5 [41.7 to 79.2] | 2146.4 [1309.0 to 3519.7] | 541.1 [31.3 to 9362.1] | 78.9 [42.6 to 146.1] | 50.0 [NA to NA] — Below level of detection
  Week 30 (N:18,6,38,20,4,6,24,5,14,3) | 3780.6 [1941.7 to 7360.9] | 477.1 [85.4 to 2664.5] | 8682.0 [5670.1 to 13293.8] | 1574.5 [568.2 to 4363.1] | 552.2 [37.8 to 8075.8] | 317.0 [27.5 to 3654.9] | 12939.5 [8634.4 to 19391.2] | 1374.9 [54.4 to 34722.9] | 1889.4 [570.8 to 6254.5] | 4360.1 [30.3 to 627361.8]
  Week 36 (N:18,6,36,20,4,9,25,5,14,3) | 2927.8 [1368.7 to 6262.8] | 267.1 [53.6 to 1331.2] | 5946.6 [3807.1 to 9288.6] | 1029.4 [346.4 to 3059.1] | 282.9 [43.5 to 1838.7] | 428.0 [83.8 to 2186.8] | 6228.9 [3794.3 to 10225.7] | 706.7 [33.6 to 14852.3] | 1018.5 [297.8 to 3483.6] | 1164.2 [23.4 to 57811.5]
  Week 50 (N:17,6,37,20,4,8,20,5,13,3) | 1843.8 [776.1 to 4380.0] | 141.3 [24.5 to 813.2] | 3146.6 [1945.8 to 5088.4] | 512.4 [176.5 to 1487.4] | 169.6 [35.8 to 804.5] | 333.6 [63.0 to 1767.0] | 2439.0 [1369.5 to 4343.8] | 527.7 [33.4 to 8348.8] | 651.3 [189.9 to 2233.5] | 401.4 [4.5 to 35461.1]
  Week 56 (N:17,6,32,19,4,8,12,4,5,3) | 4958.8 [2257.8 to 10891.0] | 1441.4 [159.3 to 13045.1] | 10412.4 [6365.4 to 17032.7] | 4562.2 [2233.3 to 9319.8] | 1720.0 [108.1 to 27356.9] | 3451.0 [478.9 to 24871.3] | 5241.2 [2459.3 to 11170.1] | 2216.1 [38.0 to 129086.9] | 578.3 [26.6 to 12559.5] | 8033.5 [584.5 to 110404.7]
  Week 66 (N:17,6,30,19,4,7,8,5,3,3) | 2765.0 [1190.8 to 6420.3] | 701.5 [86.0 to 5719.3] | 6627.7 [3946.1 to 11131.5] | 2049.2 [852.2 to 4927.5] | 891.0 [32.6 to 24385.5] | 1989.2 [152.1 to 26014.2] | 4341.1 [1677.8 to 11232.1] | 1315.8 [117.1 to 14780.6] | 968.4 [43.0 to 21784.1] | 5403.5 [171.1 to 170698.5]
  Week 76 (N:14,5,23,19,4,7,5,5,3,3) | 2802.1 [1334.8 to 5882.6] | 842.5 [107.7 to 6592.3] | 3373.8 [1763.5 to 6454.6] | 1479.9 [575.1 to 3808.2] | 628.5 [26.6 to 1478.7] | 1235.3 [116.5 to 13096.6] | 2030.7 [576.9 to 7147.4] | 875.0 [94.7 to 8083.3] | 494.1 [1.2 to 198416.2] | 2042.8 [107.4 to 38841.8]
  Week 82 (N:13,5,16,18,3,7,4,4,2,3) | 6831.1 [3436.2 to 13579.9] | 5104.3 [540.8 to 48180.8] | 12261.1 [6635.8 to 22655.2] | 5771.4 [3264.4 to 10203.5] | 2768.5 [79.0 to 97040.9] | 4779.6 [706.4 to 32339.3] | 1902.0 [35.0 to 103340.7] | 3736.1 [594.2 to 23491.3] | 1617.1 [3.0 to 868223.9] | 9922.5 [2059.8 to 47798.6]
  Week 104 (N:12,5,14,17,2,5,5,2,2,3) | 2951.6 [1259.3 to 6918.3] | 1061.0 [77.8 to 14476.0] | 6644.4 [2583.6 to 17088.1] | 1565.2 [587.2 to 4172.5] | 1128.4 [0.1 to 25253974.1] | 832.4 [56.5 to 12268.2] | 1447.6 [548.5 to 3820.9] | 3654.5 [11.3 to 1181935.3] | 321.9 [0.0 to 12636639.8] | 1340.5 [421.5 to 4263.3]

ADVERSE EVENTS:
Time Frame: Approximately 24 months, starting from Day 1, inclusive 18 months of dosing and 6 months of follow-up after the last dose.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- Active / ACC 10 µg+QS-21: Participants received 10 μg of ACC-001 and 50 μg of QS-21 or 10 μg of ACC-001 alone in the lead-in study and 10 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
- Control / ACC 10µg+QS-21: Participants received 50 μg of QS-21 or PBS in the lead-in study and 10 μg of ACC-001 and 50 μg of QS-21 in the extension study. Test article was given by intramuscular injection into the deltoid muscle at 0, 6, 12, and 18 months.
Arm/Group | ACC 3 µg+QS-21 / ACC 3 µg+QS-21 | QS-21 / ACC 3 µg+QS-21 | Active / ACC 10 µg+QS-21 | Control / ACC 10µg+QS-21 | Active / ACC 30 µg+QS-21 | Control / ACC 30 μg+QS-21
Serious Adverse Events (participants affected / at risk) | 6/21 | 0/6 | 16/65 | 2/14 | 4/33 | 4/20
Other Adverse Events (participants affected / at risk) | 19/21 | 6/6 | 55/65 | 13/14 | 23/33 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACC 3 µg+QS-21 / ACC 3 µg+QS-21 (N=21) | QS-21 / ACC 3 µg+QS-21 (N=6) | Active / ACC 10 µg+QS-21 (N=65) | Control / ACC 10µg+QS-21 (N=14) | Active / ACC 30 µg+QS-21 (N=33) | Control / ACC 30 μg+QS-21 (N=20)
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1
Cerebral haemosiderin deposition (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dementia Alzheimers type (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic mass (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Agitated depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Raynauds phenomenon (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACC 3 µg+QS-21 / ACC 3 µg+QS-21 (N=21) | QS-21 / ACC 3 µg+QS-21 (N=6) | Active / ACC 10 µg+QS-21 (N=65) | Control / ACC 10µg+QS-21 (N=14) | Active / ACC 30 µg+QS-21 (N=33) | Control / ACC 30 μg+QS-21 (N=20)
Injection site pain (General disorders) | 4 | 0 | 11 | 2 | 5 | 6
Injection site erythema (General disorders) | 4 | 0 | 5 | 1 | 5 | 4
Injection site swelling (General disorders) | 3 | 0 | 5 | 0 | 4 | 1
Fatigue (General disorders) | 2 | 1 | 4 | 0 | 1 | 0
Injection site bruising (General disorders) | 1 | 0 | 1 | 0 | 2 | 1
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 1 | 0 | 3
Injection site pruritus (General disorders) | 1 | 0 | 4 | 0 | 0 | 0
Injection site induration (General disorders) | 3 | 0 | 1 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 2 | 0 | 1 | 1
Asthenia (General disorders) | 3 | 0 | 0 | 0 | 0 | 0
Induration (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site hypersensitivity (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 4 | 9 | 1 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 6 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3 | 2 | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Infected bites (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 3 | 4 | 5 | 2 | 3 | 1
Depression (Psychiatric disorders) | 3 | 0 | 3 | 3 | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 4 | 1 | 1 | 0
Aggression (Psychiatric disorders) | 1 | 1 | 2 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 4 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Delusional perception (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 5 | 2 | 2 | 2
Headache (Nervous system disorders) | 1 | 0 | 6 | 1 | 3 | 1
Cognitive disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 2
Myoclonus (Nervous system disorders) | 1 | 1 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 2 | 0 | 0 | 0
Dementia Alzheimers type (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyperreflexia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 3 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 1 | 7 | 2 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 1 | 2 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1 | 2 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 3 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 5 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Bartonella test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Vitamin B1 decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Heterophoria (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
In 2013 the sponsor decided that ACC-001 would not be further developed in mild to moderate Alzheimer's disease, study drug administration was discontinued, and remaining participants were followed for safety for up to 6 months after last injection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.